CLINICAL TRIAL: NCT06994702
Title: Evaluation of the Impact of the MRI Restraint System on the Quality of the Synthetic Scan for Intracranial Radiotherapy Treatment: Feasibility Study
Brief Title: Impact of the MRI Restraint System on the Quality of the Synthetic Scan for Intracranial Radiotherapy Treatment
Acronym: ISTRI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ICO-2024-24
Record Dates: First submitted 2025-04-08; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Device Ineffective
Keywords: Synthetic CT; MRI
MeSH Terms: interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MRI with thermoformed masks (Experimental): MRI performed in the position of cerebral radiotherapy treatment
  Interventions: Device: MRI without mask; Device: MRI with mask 1; Device: MRI with mask 2

INTERVENTIONS:
Device: MRI without mask — MRI in position of cerebral radiotherapy treatment without mask
Device: MRI with mask 1 — MRI in position of cerebral radiotherapy treatment with mask 1
Device: MRI with mask 2 — MRI in position of cerebral radiotherapy treatment with mask 2

SUMMARY:
In radiotherapy, CT scans are the reference imaging tool for treatment planning, as they provide the electron density of the tissues required to calculate the dose. Magnetic Resonance Imaging (MRI) is used as a complement to CT to contour target volumes and organs at risk. While the properties of CT allow us to determine the electron density of tissues, the properties of MRI allow us to determine the proton density of tissues. MRI therefore provides better tissue contrast, but cannot be used directly to calculate the dose. In recent years, MRI-only protocols have been introduced to remove the need for a CT examination and avoid possible MRI-CT registration errors. Dose calculations are then performed on MRI images converted into synthetic CT images (sCT) using software based on artificial intelligence (for the most recent). Various commercial solutions are available for generating these sCTs, and the ICO already has experience of evaluating them.

While MRI scans for diagnostic purposes are performed in the free position, the generation of an sCT for treatment preparation requires the MRI scan to be performed in the radiotherapy position. For cranial lesions, a thermoformed mask fixed to the table is made for each patient. Depending on the type of treatment and its associated degree of precision, different types of mask exist at the ICO: '3-point' for normo-fractionated treatments and 'stereo' for treatments of 1 to 3 fractions. The use of these masks during the MRI examination can interfere with the correct positioning of the antennae and thus lead to a deterioration in the quality of the images obtained (MRI and, by repercussion, sCT).

The aim of this study was to evaluate the impact of the 2 thermoformed masks used at the ICO on the quality of a synthetic scan for 3 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Male > 18 years
2. Health professional practising at the ICO
3. Volunteer who has signed the consent form
4. Volunteer available to carry out the 3 MRI scans

Exclusion Criteria:

1. Claustrophobia
2. Foreign metal objects (metal splinters, filings, shotgun pellets, etc.)
3. Woman

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate quality of a synthetic scanner generated from an MRI performed in the position of cerebral radiotherapy treatment with 2 thermoformed masks | 1 day
  The quality is measured in Hounsfield Units (HU) on each of the structures outlined on the MRI scans and reproduced on the sCT scans.

SECONDARY OUTCOMES:
Comparison of the quality of MRI images with and without restraint | 1 day
  Mesure of signal-to-noise ratio (SNR)
Comparison of the quality of MRI images with and without restraint | 1 day
  Mesure of contrast-to-noise ratio (CNR)
Studying the integration of a field map into routine clinical practice | 1 day
  Measurement of acquisition
Studying the integration of a field map into routine clinical practice | 1 day
  Measurement of analysis time

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane DUFRENAIX, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (1):
- Institut de Cancerologie de L'Ouest, Angers, France

IPD SHARING:
Plan to Share IPD: No